CLINICAL TRIAL: NCT02658617
Title: Functional Neuroanatomy and Regional Metabolism Before and After Treatment With Duloxetine: A Combined fMRI and MRS Study in Major Depression
Brief Title: Functional Neuroanatomy and Regional Metabolism Before and After Treatment With Duloxetine
Status: Completed | Type: Observational
Sponsor: Heinz Boeker (Other)
Responsible Party: Sponsor-Investigator, Heinz Boeker, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: PUK09
Record Dates: First submitted 2016-01-12; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Depression
Keywords: Empathy; Interoceptive Awareness; fMRI; MRS
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: 20 patients were enrolled. Subjects were investigated with magnetic resonance spectroscopy (MRS), functional magnetic resonance imaging (fMRI) and also underwent a psychodiagnostic assessment (evaluating the severity of depression: Hamilton Depression Rating Scale and Beck Depression Inventory; measuring hopelessness: Beck Hopelessness Scale; measuring Alexithymia: Toronto Alexithymia Scale; measuring self-perception: Body Perception Questionnaire). 1-2 days after the imaging patients started the treatment with duloxetine: 30mg for the first three days, then 60-90mg.
- healthy controls: Subjects were investigated with magnetic resonance spectroscopy (MRS), functional magnetic resonance imaging (fMRI) and also underwent a psychodiagnostic assessment (evaluating the severity of depression: Hamilton Depression Rating Scale and Beck Depression Inventory; measuring hopelessness: Beck Hopelessness Scale; measuring Alexithymia: Toronto Alexithymia Scale; measuring self-perception: Body Perception Questionnaire).

SUMMARY:
The findings may guide future investigations on novel therapeutic targets in depressive subjects. Based on the depicted link between personality traits and altered brain metabolism and function, the latter might be used as supporting objective measures and possible biomarkers for increased depression risk.

DETAILED DESCRIPTION:
Interoceptive awareness (IA) is the awareness of bodily signals and has been highlighted as important in many early theories of emotion. William James was one of the first to present a psychological theory linking viscero-afferent feedback to emotional experience. The processing of bodily and thus interoceptive stimuli may be a crucial component in yielding empathy, since affective states are often assumed to involve awareness of one´s own bodily state. The assumption of a close relationship between interceptive awareness and empathy is further supported when considering the regions recruited during both processes, like the insula and the anterior cingulate cortex. Although especially the affective component may implicate interoception and interoceptive awareness, the impact of interoception on empathy has never been evaluated behaviorally or neurophysiologically.

Also associated with altered insula and anterior cingulate cortex (ACC) function is Alexithymia. Alexithymia, a personality trait, is marked by cognitive and affective features including difficulties in identifying and describing feelings as well as in distinguishing feelings from bodily sensations of emotional arousal. Recent studies found a negative correlation between prefrontal glutamate (Glu) and mental perspective taking as well as extraversion. Even though several functional imaging studies investigated the neuronal signatures of interoceptive awareness and the personality trait alexithymia, little is known about the functional relevance of neurotransmitter concentrations

ELIGIBILITY:
Inclusion Criteria:

* acute depressive episode

Exclusion Criteria:

* major medical illness
* history of seizures, head trauma with loss of consciousness
* abnormal clinical laboratory test result, and pregnancy
* atypical forms of depression
* suicidal ideation
* any additional psychiatric disorder
* history of substance abuse or dependence
* electroconvulsive therapy in the previous 6 months

Healthy subjects without any psychiatric, neurologic, or medical illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with an acute depressive episode (n = 20; 10 females; mean age ± SD age, 32.2 ± 10.3 years; number of episodes 2.7 ± 1.9; age of onset 26.7 ± 9.1 years) were recruited from the inpatient department of psychiatry at the University of Zurich. All patients were either medication naïve or not on any psychotropic medication for at least 6 weeks prior to study enrollment. Participants were entered into the study after a full explanation of the purpose of the study and the study procedures and after written consent was obtained as approved by the University of Zurich's institutional review board.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in brain activation patterns after 6 weeks treatment with duloxetine | up to 2 months